CLINICAL TRIAL: NCT02840292
Title: Effect of Maternal Hemoglobin on Neurobehavioural Development of Late Preterm Neonates : A Cohort Study
Status: Completed | Type: Observational
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, DR. VIKRAM DATTA, Professor,Department of Neonatology, Lady Hardinge Medical College
Other Study IDs: Hemoglobin and Neurobehaviour
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Anemia
Keywords: Late Preterms; Neurobehavioral Assessment of Preterm Infants (NAPI)
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cases: Late preterm neonates (>34weeks but <37weeks of gestation) with maternal hemoglobin < 11gm/dl
- Controls: Late preterm neonates (>34weeks but <37weeks of gestation) with maternal haemoglobin ≥ 11gm/dl

SUMMARY:
The study entitled 'Effect of maternal hemoglobin on neurobehavioral development of late preterm neonates' was done with an objective to determine whether low maternal hemoglobin (<11gm/dl), in late preterm neonates(>34weeks but less than 37weeks gestational age) correlates with poor neurobehavioral outcome using the Neurobehavioral Assessment of Preterm Infants(NAPI) tool, thereby allowing for earlier rehabilitative intervention to be undertaken to improve their long term outcomes and to generate useful data on a previously well recognised but under researched entity.

DETAILED DESCRIPTION:
Prevalence of anemia in India is among the highest in the world. A high proportion of women in both industrialized and developing countries become anemic during pregnancy. The major concern about the adverse effects of anemia on pregnant women and their offsprings is the belief that this population is at a greater risk of perinatal mortality and morbidity. Apart from this, it is well known that anemia per se is associated with higher incidence of premature births and low birth weight babies. Infants with iron deficiency anemia have significantly lower motor and mental scores and decreased language capabilities and body balance-coordination skills. Such infants also have a decreased learning ability. Iron deficiency anemia during the developmental stage can lead to reduced myelination of the spinal cord, as well as a change in myelin composition; abnormalities in neurotransmitters' metabolism and alteration in brain energy metabolism. The Neurobehavioral Assessments of Preterm Infants (NAPI) is a research tool to monitor the developmental progress and differential maturity of preterm infants ranging between 32weeks and 37weeks (full term). This test is used to identify persistent lags in development, as a research tool to assess effects of interventions and to study individual differences and basic developmental questions. The reliability and clinical validity of this test has been thoroughly investigated and normative data has been established.

Objective - To evaluate the neurobehavioral development at 37weeks of post conceptional age in late preterm infants born to mothers with hemoglobin <11gm/dl; by a standardised scale - Neurobehavioral Assessment of Preterm Infants (NAPI).

ELIGIBILITY:
Inclusion Criteria:

* Late preterm infants born to mothers <35yrs of age and born between 34weeks to 36.6weeks of gestation as calculated by last menstrual period/1st trimester ultrasound
* Clinically stable from respiratory, hemodynamic and metabolic point of view
* After receiving full, free, voluntary, informed consent from parents/family members within 24 hours of delivery.

Exclusion Criteria:

* Chorioamnionitis in pregnancy.
* Congenital malformations (antenatally diagnosed or evident on clinical examination)
* Neonates admitted to NICU
* Neonates requiring ventilator support
* Neonates with any neurological impairment (IVH etc)
* Neonates undergoing surgery
* Neonates with birth asphyxia
* Neonates with birth trauma
* Confirmed history of substance abuse in mother.

Ages: 34 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 100 late preterms (56 cases vs. 44 controls) fulfilling the criteria were enrolled from Main Labor Room, Maternity Ward, Operation Theatre or Post Natal Wards of the Department of Obstetrics and Gynaecology, Lady Hardinge Medical College.
  NAPI was administerd to 63 neonates (32 cases vs 31 controls).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of neurobehavioral development | 2 months
  The two sub domains of Neurobehavioral Assessment of Preterm Infants (NAPI) i.e. Motor Development and Vigor (MDV) and Alertness and Orientations (AO) were tested to evaluate the neurobehavioral development at 37weeks of post conceptional age in late preterm neonates

SECONDARY OUTCOMES:
Comparison of NAPI Score | 1 month
  The scores of the two sub domains of Neurobehavioral Assessment of Preterm Infants (NAPI) i.e. Motor Development and Vigor (MDV) and Alertness and Orientations (AO) were compared to determine the level of maturity in the neurobehavioral development in cases and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Vikram Datta, MD, DNB, Study Chair — Lady Hardinge Medical College; Dr. Sanya Chandna, MBBS, Principal Investigator — Lady Hardinge Medical College
Locations (1):
- Lady Hardinge Medical College, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided